CLINICAL TRIAL: NCT03008044
Title: Evaluation of a Percutaneous Optical Fibre Glucose Sensor (FiberSense) Across the Glycemic Range With Rapid Glucose Excursions Using the Glucose Clamp
Brief Title: Evaluation of a Percutaneous Optical Fibre Glucose Sensor (FiberSense System)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: P-4.4-C-01
Record Dates: First submitted 2016-12-16; First posted 2017-01-02 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: For the first 10 subjects, all sensors will be removed after the end of the clamp measurement day.
  The last 2 subjects will continue to wear the three sensors after the clamp study. The second clamp study will take place at Day 7±1. After the second clamp study, the commercial CGM sensor will be removed. The two FiberSense sensors will be worn for up to Day 14.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Device: FiberSense system (Experimental): 10 subjects will wear 2 FiberSense system in abdomen and upper arm respectively and Dexcom G4 Platinum CGM sensor for 1 day.
  Interventions: Device: FiberSense system
- Extension Phase (Experimental): 2 subjects will extend the wearing of the sensors up to 14 days (2 FiberSense systems to Day 14 and Dexcom sensor to Day 7±1) after the glucose clamp study.
  Interventions: Device: FiberSense system

INTERVENTIONS:
Device: FiberSense system — A novel CGM system based on a FiberSense system placed through the dermis of the patient.

SUMMARY:
This is a single center prospective study. The purpose of this study is to assess the performance of FiberSense system across the glucose measurement ranges (from hypoglycemia to hyperglycemia) as compared with a gold standard reference laboratory method (YSI glucose) in healthy volunteers.

DETAILED DESCRIPTION:
The FiberSense system is intended to be used by diabetic patients in a home use setting as a CGM system using the interstitial fluid (ISF) glucose as an indicator of blood glucose levels.The purpose of this study is to assess the performance of FiberSense system across the glucose measurement ranges (from hypoglycemia to hyperglycemia) as compared with a gold standard reference laboratory method (YSI glucose) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 18 years old.
* Nondiabetic subjects with normal fasting plasma glucose and HbA1c (≤5.6%)
* Women who are not pregnant, lactating or planning a pregnancy during their participation in the clinical study.
* Willingness, ability and commitment to comply with the testing, procedure and follow-up outlined in this protocol including (but not limited to) frequency of clinic visits and use of pre-specified glucose monitoring devices.
* Willingness to abstain from bathing and swimming during their participation in the measurement phase.
* In the opinion of the investigator, absence of any physical limitations, addictive diseases, or underlying medical conditions (including mental health) that may preclude the patient from being a good study candidate.
* Written informed consent to participate in the study provided by the patient.

Exclusion Criteria:

* Currently pregnant, as demonstrated by a positive pregnancy test at screening and on day of first sensor insertion
* Impaired hepatic function measured as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ three times the upper reference limit.
* Impaired renal function measured as serum creatinine > 1.2 times above the upper limit of normal.
* Any active acute or chronic disease or condition that, in the opinion of the investigator, might interfere with the performance of this study.
* Any active acute or chronic infectious disease that, in the opinion of the investigator, would pose an excessive risk to study staff.
* Current use or recent exposure to any medication that in the opinion of the investigator could have an influence on the patient's ability to participate in this study or on the performance of the test device.
* Extensive skin changes/diseases that preclude wearing the required number of devices on normal skin at the proposed application sites (e.g., extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis).
* Have a known allergy to medical-grade adhesives, or known hypersensitivity to any of the products used in the study.
* Known current or recent alcohol or drug abuse
* Blood donation of more than 500 ml within the last three months
* Currently participating in another investigational study protocol where the testing or results may interfere with study compliance, diagnostic results, or data collection.
* History of epilepsy
* History of cardiac arrhythmias
* Clinically significant abnormality on ECG at screening
* An identified protected vulnerable patient (including but not limited to those in detention, or a prisoner).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-08; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Overall performance of the FiberSense device as compared with YSI | 1 day
  Proportion of FiberSense readings within ≤15% of the reference (YSI) reading for blood glucose levels >100 mg/dl (5.55 mmol/l), and the proportion of FiberSense readings within ≤15 mg/dl (0.83 mmol/l) of the YSI reading for blood glucose levels ≤100 mg/dl.

SECONDARY OUTCOMES:
Mean relative differences in FiberSense measured glucose from the reference laboratory standard (YSI) | 1 day
Mean Absolute Relative Differences in FiberSense measured glucose from the reference laboratory method (YSI) | 1 day
Accuracy of glucose rate of change measured by FiberSense sensor compared to glucose rate of change measured using the reference laboratory method (YSI) | 1 day
Lag time between FiberSense readings and reference laboratory method (YSI) results during induced glucose excursions | 1 day
Precision of FiberSense system readings: Precision Absolute Relative Differences with comparison of FiberSense system locations (inter and intra) | 1 day
Percentage of readings that are within 15% of the YSI values | 1 day
  Comparisons of the percentage of readings from Dexcom and Fibersense, and comparisons of the percentage of readings from Bayer Contour Next and Fibersense, will be done separately during analysis.
Percentage of readings that are within 20% of the YSI values | 1 day
  Comparisons of the percentage of readings from Dexcom and Fibersense, and comparisons of the percentage of readings from Bayer Contour Next and Fibersense, will be done separately during analysis.
Percentage of readings that are within 30% of the YSI values | 1 day
  Comparisons of the percentage of readings from Dexcom and Fibersense, and comparisons of the percentage of readings from Bayer Contour Next and Fibersense, will be done separately during analysis.
Percentage of readings that are within 40% of the YSI values | 1 day
  Comparisons of the percentage of readings from Dexcom and Fibersense, and comparisons of the percentage of readings from Bayer Contour Next and Fibersense, will be done separately during analysis.
Percentage of readings that are greater than 40% of the YSI values | 1 day
  Comparisons of the percentage of readings from Dexcom and Fibersense, and comparisons of the percentage of readings from Bayer Contour Next and Fibersense, will be done separately during analysis.
Adverse Event Reporting | 14 days
Median relative differences in FiberSense measured glucose from the reference laboratory standard (YSI) | 1 day
Median Absolute Relative Differences in FiberSense measured glucose from the reference laboratory method (YSI) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Chow, Dr., Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No